CLINICAL TRIAL: NCT01430780
Title: A Prospective Study to Evaluate the Influence of Oxygen Free Radical Injury Induced by Long-term Nitrates Therapy on Vasodilation Function of Patients With Coronary Heart Disease
Brief Title: A Prospective Study to Evaluate the Effect of Chronic Nitrate Therapy on Vasodilation Function in Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiangtao Lai, MD, Zhejiang University
Other Study IDs: 2009A062
Record Dates: First submitted 2011-09-01; First posted 2011-09-08 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; nitrate; endothelium
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: placebo
  Interventions: Drug: control group
- nitrate group: Isosorbide Mononitrate orally 20mg twice per day.
  Interventions: Drug: nitrate group

INTERVENTIONS:
Drug: nitrate group — Isosorbide Mononitrate orally 20mg twice per day.
  Groups: nitrate group
Drug: control group — placebo
  Groups: control group

SUMMARY:
Basic studies has showed that sustained use of nitrates might associated with adverse effects on vascular function mediated by an increase in nitrate-induced oxidative stress. But it remains unclear whether oxidative stress increases with endothelial function impairment in patients with coronary artery disease (CAD) during administration of long-term oral nitrates. The investigators evaluated whether administration of long-term isosorbide mononitrate (ISMN) treatment was associated with oxidative stress increase and endothelial function impairment in patients with CAD.

DETAILED DESCRIPTION:
Organic nitrates are widely prescribed for the treatment of angina pectoris in patients with coronary artery disease (CAD). In China, many patients with CAD are prescribed nitrates as a long-term treatment. The most commonly prescribed nitrates for long-time treatment is isosorbide mononitrate (ISMN). The reason for their use is that the majority of physicians believe chronic therapy with organic nitrates is associated with an improvement in symptoms and has neutral or potentially beneficial effects on long-term patient outcome, although this assumption remains unproven.

Recently, multiple lines of evidence documented that sustained use of nitrates was associated with adverse effects on vascular function which appeared to be mediated by an increase in nitrate-induced oxidative stress. The accumulation of oxygen free radicals during chronic nitrate therapy was associated with endothelial dysfunction, increased arterial sensitivity to vasoconstrictors and the development of abnormalities in a number of important enzymes involved in the regulation of vascular homeostasis, including the superoxide dismutase, protein kinase C, matrix metalloproteinases, and prostaglandin synthase. This may lead to development of nitrate tolerance, endothelial dysfunction. Furthermore, endothelial dysfunction is a risk factor for worse prognosis of patients with CAD.

Up to date, some clinical research focus on how to prevent tolerance and clinical outcome of nitrate therapy were involved short follow-up periods of only a few weeks. It is too short to assess the true clinical impact of nitrate-induced endothelial dysfunction, and the safety of long-term nitrate therapy requires systematic review. So prospective, randomized study with longer treatment period is needed to observe the chronic impact of nitrate therapy on endothelial function.

Therefore, the investigators prospectively investigated whether long-term ISMN therapy had any influence on endothelial function evaluated by brachial artery ultrasound imaging during reactive hyperemia in patients with catheterization confirmed CAD, and whether this was associated with increased oxidization or inflammation burden.

ELIGIBILITY:
Inclusion Criteria:

* Individuals were considered eligible for enrollment if they had at least 1 significant de novo stenosis (reduction ≥50% of the lumen diameter) on any coronary vessel at angiography.

Exclusion Criteria:

* Patients with liver and renal failure with creatinine>3 mg/dL were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with catheterization confirmed coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
flow-mediated dilation | one year
  Endothelial function evaluated by brachial artery ultrasound imaging during reactive hyperemia.

SECONDARY OUTCOMES:
serum superoxide dismutase (SOD) level | one year
  Superoxide dismutase (SOD) was determined by Xanthinoxidase method.
serum malondialdehyde (MDA) level | one year
  Malondialdehyde (MDA) was determined by thiobarbituric acid method.
serum hypersensitive C-reactive protein (hsCRP) level | one year
  An ELISA was used to determine hypersensitive C-reactive protein (hsCRP).

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Lai, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- Department of Cardiology, First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Lai J, Wu B, Sun J, Shang Y, Zhu J. Long-term isosorbide mononitrate treatment impairs endothelial function in patients with coronary artery disease. Coron Artery Dis. 2013 Nov;24(7):566-71. doi: 10.1097/MCA.0000000000000029. PMID 23994882